CLINICAL TRIAL: NCT04561934
Title: Clinical and Radiographic Evaluation of Deep Occlusal Carious Molars Treated With Partial Caries Removal With and Without Using Silver Diamine Fluoride (SDF) Prior to Resin Composite Restoration. (A Randomized Clinical Trial)
Brief Title: Clinical and Radiographic Evaluation of Deep Occlusal Carious Molars Treated With Partial Caries Removal With and Without Using Silver Diamine Fluoride (SDF) Prior to Resin Composite Restoration.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Laila Akmal Emad Eldien Elokaly, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2629
Record Dates: First submitted 2020-09-20; First posted 2020-09-24 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Partial Caries Removal
MeSH Terms: interventions — silver diamine fluoride

STUDY DESIGN:
Intervention Model Description: eighty teeth are assigning into two equal groups of forty
Who Masked: Participant, Outcomes Assessor
Masking Description: The operator cannot be blinded because of the difference in operative and application procedures between control and intervention groups. The operator will blind until randomization into groups to avoid bias regarding the application of SDF to which tooth. However, the patients and assessors who carried out the radiographic assessment will be blinded of the treatment group. Finally, the treatment results will assess blindly by a statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- resin modified glassionomer cement (Experimental): Application of Resin modified glass ionomer cement (RMGIC) (Fuji Lining LC; GC, Tokyo, Japan) prior resin composite restoration (Filtek Z350 XT,3MESPE)
  Interventions: Other: resin modified glassionomer cement
- silver diamine flouride (Active Comparator): Application of 38% SDF (Riva Star, SDI, Bayswater, Australia), and Resin modified glass ionomer cement (RMGIC) (Fuji Lining LC; GC, Tokyo, Japan) prior resin composite restoration (Filtek Z350 XT,3MESPE).
  Interventions: Drug: Silver diamine fluoride

INTERVENTIONS:
Drug: Silver diamine fluoride — Application of 38% SDF (Riva Star, SDI, Bayswater, Australia), and Resin modified glass ionomer cement (RMGIC) (Fuji Lining LC; GC, Tokyo, Japan) prior resin composite restoration (Filtek Z350 XT,3MESPE).
  Arms: silver diamine flouride
Other: resin modified glassionomer cement — resin modified glassionomer cement
  Arms: resin modified glassionomer cement

SUMMARY:
The aim of the study is to evaluate the effect of SDF in maintaining pulp health after partial caries removal in permanent teeth with deep occlusal carious lesion clinically and radiographically

DETAILED DESCRIPTION:
Pre-operative clinical assessment:

Before starting the study, the participants will undergo radiographic examination to ensure that the carious lesion penetrate at least the inner one-half of the dentin thickness and show normal lamina dura and periodontal ligament.

Cavity preparation procedure:

Under local anesthesia and rubber dam isolation. A high-speed handpiece (T3 mini, Sirona GmbH, Bensheim, Germany) under air/water coolant and No. #245 bur will use to obtain the cavity outline allowing access to the carious lesion beyond the dentin-enamel junction. (Bitello-Firmino et al., 2018). Then, complete caries excavation will be performed in the cavity except at the floor where partial caries removal will be performed using sharp sterile excavator. Then cavities will be randomly divided into two groups according to the selected sealed envelopes.

Restorative treatment:

* For the control group Isolation of the prepared cavity will be maintained using rubber dam. The cavity will be lined with a liquid-paste, resin-modified GIC liner (Fuji Lining LC Paste Pak; GC, Tokyo, Japan) in 0.5-1 mm thickness over the entire dentin floor, and then bonded with self-etching adhesive (Clearfil SE Bond; Kuraray Medical, Okayama, Japan).The bonded cavity will be filled incrementally with resin composite restoration (Filtek Z350 XT,3MESPE) and then will be light cured for 20s.
* For the intervention group Isolation of the prepared cavity will be maintained using rubber dam. Riva star SDF will be applied over the entire dentin floor in two steps: The first Step, the silver capsule solution will be applied using the silver brush provided. Then the second Step, the green capsule solution will be applied in a generous amount immediately after applying the silver capsule solution at the same treated site until the treated surface color change from creamy white to clear. And then, after one-minute Riva star SDF will be blot dried or if the clinical situation permits, will be wash thoroughly with water for at least 10 seconds and then air dry without desiccation. Resin modified glass-ionomer liner will be then applied over Riva star SDF prior to resin composite restoration application.

  12. Outcomes: The primary outcome of this clinical trial is success, express as a binary variable indicating whether the restored tooth maintained its pulp vitality after 12 months (T2). Success will evaluate by a positive response to cold pulp testing, absence of spontaneous pain, no tenderness to percussion, absence of periapical radiolucency .

ELIGIBILITY:
Inclusion Criteria:

* Class I carious lesions.

  * Lower and upper molars.
  * 18 -50 years.
  * Not received antibiotic therapy since 1 month before sampling.
  * Males or Females (Both genders).
  * Co-operative patients approving the trial

Exclusion Criteria:

* • known allergic reaction to fluoride or silver

  * Systemic disease or severe medical complications.
  * Periodontal problem.
  * Mobile teeth, arrest caries and non-vital teeth
  * Ulcerative gingivitis, and Stomatitis.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
clinical survival | 12 months
  express as a binary variable indicating whether the restored tooth maintained its pulp vitality

IPD SHARING:
Plan to Share IPD: Undecided